CLINICAL TRIAL: NCT05788198
Title: Integrated Depression Care Project
Brief Title: Integrated Depression Care
Acronym: IDECA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Universiteit Antwerpen (Other); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NOPRODDEP4002
Record Dates: First submitted 2021-11-19; First posted 2023-03-28 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Depression Mild; Depression Moderate; Depression Severe
MeSH Terms: interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Intervention Model Description: Pre/Posttest implementation study.
Masking Description: Investigators, care providers, and participants will know treatment arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated care arm (Experimental): Case management in primary care setting (integration at general practitioners' practices), Depression and population management education for general practitioners, shared care guidance protocol including a medication path (drug classes, no specific drugs specified, based on available depression guidelines in Belgium).
  Interventions: Other: Integrated care

INTERVENTIONS:
Other: Integrated care — The intervention will be modelled based on the most frequently reported patient, family physician and specialist barriers in depression management. In this project, multiple interventions aiming to tackle these barriers will be set up, with the WHO Framework on Integrated People-Centred Health Services (IPCHS) serving as conceptual backbone to the study (Table 1). The IPCHS distinguishes five interdependent strategies supporting a shift in healthcare delivery, management and funding towards universal health coverage. These strategies are:
  1. empowering and engaging people and communities;
  2. strengthening governance and accountability;
  3. reorienting the model of care;
  4. coordinating services within and across sectors;
  5. creating an enabling environment.

SUMMARY:
The Integrated DEpression CAre (IDECA) Programme is a multi-faceted intervention strategy aiming to improve guideline adherence and shared care practices for depression management in both providers and patients, as measured through a set of process and clinical outcome indicators (primary outcome measure).

DETAILED DESCRIPTION:
The following deliverables apply:

1. Development and implementation of a shared care protocol for depression management involving primary, secondary and tertiary care levels;
2. Training module for physicians and other care providers in population health management for patients with depression;
3. Training module for case managers/integration of a case management function into existing depression service offerings;
4. A patient education module for depression self-management;
5. A financing model for integrated depression care.

ELIGIBILITY:
Inclusion Criteria:

* persons between 18-65
* presenting to the general practitioner's office
* with depressive symtomatology

Exclusion Criteria:

* Severe depression warranting direct referral to specialized services

Inclusion criteria are kept broad on purpose as it's one of the research questions to define for which patients the intervention (namely the case management) is appropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intervention integration | 14 months
  Nomad questionnaire (4 monthly), followed by focus groups following Balint method, and individual interviews.

SECONDARY OUTCOMES:
Depression | 12 months
  PHQ-9 (Patient Health Questionnaire. DSM-5 depression), A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression
Depression and anxiety | 12 months
  OQ-45-2 (Outcome Questionnaire. Transdiagnostical instrument focused on anxiety and depression) Total Score
  * Total scores (≥ 64) reflect increased distress
    * High is anything above 105
    * Moderately High is between 83 and 105
    * Moderate is between 64 and 82
    * Low is anything below 64 Symptom Distress (SD)
  * Scores (≥ 37) indicate subjective discomfort Interpersonal Relations (IR)
  * Scores (≥ 16) reflect problems in interpersonal relations. Social Role (SR)
  * Scores (≥ 13) indicate dissatisfaction, conflict, distress, and inadequacy in performance of tasks related to employment, school, family roles and leisure life.
Medication adherence and self-efficacy | 12 months
  MARS-5 (Medication adherence report score) Each item was rated on a 5-point Likert scale, and the range of the MARS-5 total score is between 5 and 25. A higher score on the MARS-5 represents better medication adherence. <21 suboptimal adherence.
  MUSE (Medication Understanding and Use Self-Efficacy Scale). Score 8-32. Higher scores are better.
Resource use | 12 months
  iMCQ (The iMTA Medical Consumption Questionnaire) to capture depression-related resource use
Health-related Quality of Life | 12 months
  EQ5D5L (EuroQol 5 Dimensions 5 levels). Score 0 equals death and 1 perfect health.
Health literacy | 12 months
  HLS-EU-Q16. Considering the HLS-EUQ16 score, three levels of health literacy were defined: - inadequate HL (0-8) - problematic HL (9-12) - adequate HL (13-16)

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Borgermans, PhD, Principal Investigator — University Ghent; Lieven Annemans, PhD, Study Chair — University Ghent
Locations (2):
- Belgium (2):
  - ELZ Mechelen-Katelijne, Mechelen
  - ELZ Voorkempen, Zoersel

IPD SHARING:
Plan to Share IPD: No
None, except anonymized data for peer review.